CLINICAL TRIAL: NCT04635813
Title: The Impact of COVID-19 Pandemic on Thyroid Surgery in Italy: Results From a Nation-wide Multicentric Study
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Assistant Professor, University of Cagliari
Other Study IDs: THYCOVIT
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - COVID group: Patients that underwent surgery during COVID-19 pandemic
  Interventions: Procedure: Thyroidectomy
- Group 2 - control group: Patients that underwent surgery during 2019
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Thyroidectomy

SUMMARY:
Italy has been on the frontline of the COVID-19 pandemic, caused by the coronavirus SARS-CoV-2, the need to focus resources to deal with the pandemic led to a disruption of routine surgical care, as well as activity for oncologic and chronic disease. The aim of this study was to evaluate the impact of COVID-19 pandemic on surgical activity of the Italian Units of Endocrine Surgery belonging to the SIUEC (Italian Society of Endocrine Surgery), the most important national scientific society of endocrine surgery.The aim of this study was to evaluate the impact of COVID-19 pandemic on surgical activity of the Italian Units of Endocrine Surgery belonging to the SIUEC (Italian Society of Endocrine Surgery), the most important national scientific society of endocrine surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients that had undergone thyroidectomy during COVID-19 pandemic (from the 9th March to the 31st August 2020), defined as case group, or during the same period of the previous year (from the 9th Match to the 31st August 2019), defined as control group.

Exclusion Criteria:

* incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thyroid disease
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Quantify the overall reduction of surgical activity for thyroid disease | 1 year

SECONDARY OUTCOMES:
Quantify if the number of thyroid cancers operated during COVID-19 pandemic was significant different from the number of patients operated during the same period of the previous year | 1 year
Quantify the number of aggressive tumors operated during COVID-19 pandemic and the same period of the previous year | 1 year
  Comparison between the number of patients operated during COVID-19 pandemic with aggressive thyroid carcinoma (with lymph node metastasis, and/or extrathyroidal extension, and/or multifocality) with patients with aggressive thyroid carcinoma operated during the same period of the previous year

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No